CLINICAL TRIAL: NCT05897645
Title: High-resolution Magnetic Resonance Imaging of Intracranial Atherosclerotic Plaques in Ischemic Stroke (HRMRI-ICAS): a Prospective, Multicenter Cohort Study
Brief Title: High-resolution Magnetic Resonance Imaging of Intracranial Atherosclerotic Plaques in Ischemic Stroke
Status: Recruiting | Type: Observational
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, chief, General Hospital of Shenyang Military Region
Other Study IDs: Y(2022)070
Record Dates: First submitted 2023-05-23; First posted 2023-06-09 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Stroke; Intracranial Atherosclerosis; High Resolution Magnetic Resonance Imaging
MeSH Terms: conditions — Stroke; Intracranial Arteriosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Registration — collect clinical date, assess the morphologic characteristics of plaque

SUMMARY:
Intracranial atherosclerotic disease is the most common cause of ischemic stroke in Asia, also in China. Currently, despite vascular recanalization therapy, statins are one of the main drug choices for treating atherosclerotic plaque. High resolution magnetic resonance imaging (HRMRI) can accurately assess the status of intracranial and extracranial arterial plaque, and has high consistency with histopathology. Thus, HRMRI technology has been widely used to monitor the efficacy of drug treatment for atherosclerotic plaque in clinical trials or practice.

As a non-invasive technique, HRMRI make it possible to assess the morphologic characteristics of vascular wall and plaque composition of intracranial artery in vivo. It can quantitative analysis including components such as lipid-rich necrotic core, fiber cap thickness, intra-plaque hemorrhage, calcification, etc. Therefore, it is crucial for evaluating the etiology of ischemic stroke and developing secondary prevention strategies.

At present, there is a lack of large-scale and prospective study to evaluate the etiology of ischemic stroke including cryptogenic stroke based on HRMRI. In this context, this study aims to establish a multi center HRMRI database of intracranial arteries among Chinese patients with ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient age ≥40 years
* 2. Time of stroke onset: within 2 week
* 3. Baseline NIHSS score ≤16
* 4. Ischemic stroke confirmed by head CT or MRI
* 5. Premorbid mRS ≤1
* 6. The degree of stenosis of extracranial arteries including internal carotid artery, vertebral artery on the lesion side ≤50%
* 7. The culprit plaque or possible culprit plaque with plaque burden of 40% or more found by HRMRI in the proximal part of the middle cerebral artery M1 segment or basilar artery of ipsilateral lesion
* 8. Signed informed consent

Exclusion Criteria:

* 1. Intracranial hemorrhage found by head CT
* 2. Had a contraindication to MRI,or could not complete required MRI sequences
* 3. Intracranial tumor, arteriovenous malformation, or aneurysm
* 4. Comorbidity with any serious diseases and life expectancy is less than one year
* 5. Pregnancy
* 6. Patients not suitable for this clinical studies considered by researcher

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with ischemic stroke who performed HRMRI
Sampling Method: Probability Sample
Enrollment: 2110 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence of stroke | 360 days
  including ischemic or hemorrhagic stroke

SECONDARY OUTCOMES:
Recurrence of stroke | 90 days, 180 days
  including ischemic or hemorrhagic stroke
the composite events of cardiovascular events | 90 days, 180 days, 360 days
  Cardiovascular events include cardiovascular death, stroke, non-fatal myocardial infarction, and arterial revascularization
distribution of modified Rankin Scale (mRS) score | 90 days, 180 days 360 days
  mRS score range from 0 to 6: 0 [no symptoms] to 6 [death]
The relationship between characteristics of intracranial plaques and functional independence | 90 days, 180 days, 360 days
  characteristics of intracranial plaques includes plaque composition, location and morphology; functional independence is defined as modified Rankin Scale (mRS) score 0-1 (mRS score range from 0 to 6: 0 [no symptoms] to 6 [death])
The relationship between burden of cerebral small vessel disease and functional independence | 90 days, 180 days, 360 days
  burden of cerebral small vessel disease ranges from 0 to 4, with higher scores indicating greater burden; functional independence is defined as modified Rankin Scale (mRS) score 0-1 (mRS score range from 0 to 6: 0 [no symptoms] to 6 [death])

CONTACTS AND LOCATIONS:
Overall Officials: HuiSheng Chen, Principal Investigator — General Hospital of Northern Theatre Command
Locations (1):
- Department of Neurology, General Hospital of Northern Theater Command, Shenyang, China